CLINICAL TRIAL: NCT05836857
Title: The Use of Cannabis (Marijuana) and Cannabidiol (CBD) Among Cancer Patients: A Pilot Study
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0049; NCI-2023-03440 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — nabiximols; Cannabidiol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cannabis (Marijuana) and Cannabidiol (CBD): This is a survey to determine the number of cancer pain patients who use and/or used Marijuana and/or CBD for pain or other symptom burdens.
  Interventions: Behavioral: Cannabis (Marijuana); Behavioral: Cannabidiol (CBD)

INTERVENTIONS:
Behavioral: Cannabis (Marijuana) — The level of interest in learning more about cannabis for cancer pain, we can better facilitate a patient-centered approach to comprehensive treatment plans through patient education.
Behavioral: Cannabidiol (CBD) — The level of interest in learning more about cannabis for cancer pain, we can better facilitate a patient-centered approach to comprehensive treatment plans through patient education

SUMMARY:
To collect information about how patients in the pain management clinic use cannabis/CBD, including how often it is used, why it is used (for example, to manage pain or other symptoms), and where patients get their information on cannabis/CBD for pain management

DETAILED DESCRIPTION:
Objectives

Primary Objective:

The primary objective of this study is to investigate the prevalence of current and prior cannabis and/or CBD use in cancer patients who present to the pain management clinic at MDACC.

Secondary Objectives:

The secondary objective is to investigate the reason for cannabis/CBD use (e.g. pain, neuropsychiatric symptoms, recreational or other use), degree of symptom improvement with use, frequency of use, methods of use (e.g. inhaled vs. ingested), sources of information on cannabis/CBD, and patient interest in learning more from their physicians about cannabis/CBD for cancer pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Cancer patients who present to the MD Anderson Pain Medicine Clinic as a new patient or consult
3. Willing to give informed consent
4. Willing to complete the survey

Exclusion Criteria:

1. Refusal of informed consent
2. Refusal to complete the survey
3. Patients who previously completed the survey
4. Patients who opt-out or change their mind after agreeing to participate
5. Already an established patient at MDACC Pain Medicine Clinic
6. Patients scheduled to see Dr Abdi (PI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: M D Anderson Cancer Center
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Cannabis (Marijuana) and CBD (Cannabidiol for Cancer Pain Survey | through study completion; an average of 1 year.
  Score scale ranges from 1-5, Extremely interested(1),Not Interested (5)

CONTACTS AND LOCATIONS:
Overall Officials: Salahadin Abdi, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org